CLINICAL TRIAL: NCT01722682
Title: Bone Marrow vs Liver as Site for Islet Transplantation in Patients With Type 1 Diabetes: Pilot Study to Evaluate Efficacy
Brief Title: Bone Marrow vs Liver as Site for Islet Transplantation
Acronym: IsletBOM2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Piemonti Lorenzo, Head of Beta Cell Biology Unit, CO-Director Human Islet Transplantation Program (ITP), Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IsletBOM2
Record Dates: First submitted 2012-10-31; First posted 2012-11-07 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: intraportal islet infusion (Active Comparator): Patients will received islet into the liver through the portal venous circulation (standard procedure)
  Interventions: Biological: Human pancreatic islet transplantation
- B: intra BM islet infusion (Experimental): Patients will received an intra BM islet infusion at the level of the iliac crest. The direct intra BM administration will be performed following the same procedures that our institution utilizes for administration of cord-blood cells in patients with acute leukemia (Lancet Oncol. 2008;9:831). The procedure is easy and reproducible: a standard needle for BM aspiration is inserted in the iliac crest and cells are gently infused.
  Interventions: Biological: Human pancreatic islet transplantation

INTERVENTIONS:
Biological: Human pancreatic islet transplantation

SUMMARY:
The goal of this study is to evaluate safety and efficacy of bone marrow (BM) as site for pancreatic islet transplantationin humans. Our hypothesis is that BM represents a better site than liver (currently the location of choice for this procedure) thanks to its potential capacity to favor islet engraftment. To address our hypothesis we propose herein a randomized phase II trial to compare BM and liver as sites for islet transplantation in T1D patients.

DETAILED DESCRIPTION:
The study is a phase II, single center, open label, pilot study. We will recruit 12 patients with T1D to be randomly (1:1) assigned to receive islet either into the liver through the portal venous circulation (standard procedure; arm A, n=6) or directly into the BM at the level of the iliac crest (arm B, n=6). Patients will be selected from those eligible for islet Tx based on local practice and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients eligible for pancreatic islet transplantation based on local accepted practice and guidelines. This includes at least: a)clinical history compatible with T1D with insulin-dependence for >5 years; b) undetectable stimulated (arginine or MMTT) C-peptide levels (<0.3 ng/mL) in the 12 months before transplant c)presence of severe hypoglycaemic events

Exclusion Criteria:

* presence of hematologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insulin secretion under stimulation | month 12 post-Tx
  basal and -10 to 120 min time course of glucose, C-pep levels and insulin derived from the mixed meal tolerance test

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AE) and Serious Adverse Events (SAE) | throughout the study up to 1 year after first transplant
Insulin requirement | month 1, 3, 6, 9, 12 post- transplant
  Change in average daily insulin requirements
Islet function | month 1, 3, 6, 9, 12 post-Tx
  change in HbA1c, Transplant Estimated Function (TEF) and fasting C-peptide levels

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Result] Maffi P, Nano R, Monti P, Melzi R, Sordi V, Mercalli A, Pellegrini S, Ponzoni M, Peccatori J, Messina C, Nocco A, Cardillo M, Scavini M, Magistretti P, Doglioni C, Ciceri F, Bloem SJ, Roep BO, Secchi A, Piemonti L. Islet Allotransplantation in the Bone Marrow of Patients With Type 1 Diabetes: A Pilot Randomized Trial. Transplantation. 2019 Apr;103(4):839-851. doi: 10.1097/TP.0000000000002416. PMID 30130323
- See also: Related Info — http://www.hsr.it/ricerca/divisioni-centri-istituti-e-programmi-di-ricerca/islet-trasplantation-program-itp/